CLINICAL TRIAL: NCT02085564
Title: Significance of Peritoneal Washing Cytology Before and After Neoadjuvant Chemotherapy in Patients With Esophagogastric-junction Cancer
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Danish Cancer Society (Other)
Responsible Party: Principal Investigator, Rune Broni Strandby, Junior researcher, Rigshospitalet, Denmark
Other Study IDs: 050314-Rstrandby1
Record Dates: First submitted 2014-03-11; First posted 2014-03-13 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Gastroesophageal-junction Cancer
Keywords: Gastroesophageal-junction cancer; neoadjuvant chemotherapy
MeSH Terms: interventions — Peritoneal Lavage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 100ml of peritoneal washings will be obtained pr. patients x 2. The first at the staging laparoscopy, and the second initially before esophagectomy. The specimen will be analyzed for any malignant cancer cells by an authorized pathologist. Afterwards, the specimen will be destroyed.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- GEJ-cancer patients consideres resectable: All patients have biopsy verified GEJ-cancer, and has been considered for intend curative resection by a multidisciplinary panel of specialists.
  Interventions: Procedure: Peritoneal washing cytology

INTERVENTIONS:
Procedure: Peritoneal washing cytology — The methode is describes in the detailed study description
  Other Names: Peritoneal lavage

SUMMARY:
Background:

The prevalence of gastroesophageal-junction cancer (cancer between the distal part of the oesophagus, and proximal part of the stomach/GEJ-cancer) is increasing in Denmark with more than 400 patients per year. The 5-year overall survival is less than 10% for the 2/3 of the patients, which are not considered resectable. Even for the 1/3, which is treated with surgical intervention and neoadjuvant chemotherapy the overall-survival is approximately 30%.

The current Danish intended curative treatment consists of esophagectomy (surgical resection of the oesophagus with extended lymphadenectomy in abdomen and thorax (removal of lymphnodes)). Furthermore, perioperative chemotherapy consists of 6 series neoadjuvant chemotherapy (3 series before, and 3 series after operation).

Unresectable patients receive palliative chemotherapy and no resection. Peritoneal washing cytology (PWC) is a recommended prediagnostic modality in gastric cancer patients. The method is used to detect free peritoneal cancer cells in the abdominal cavity even when macroscopic carcinomatosis is not present (i.e. the cancer has spread to other parts of the abdomen).

Carcinomatosis can be found in up to 19% in gastric cancer patients often in the peritoneum. Positive peritoneal cytology (C1) can be identified in up to 7% of gastric cancer patients without metastases (C1M0), i.e. malignant cells can be identified in the peritoneal washing, but tumor spread has not been identified.

Lots of studies indicate that C1-disease is an independent prognostic predictor for decreased survival, and increased recurrence rate, comparable with M1 patients (i.e. patients with distant metastases).

The American Joint Committee on cancer recommends that C1 patients should be treated non-surgically - even when M1 disease has not been identified.

On the basis of the above, PWC can be used to identify patients at greater risk for recurrence, and thereby not candidates for intended curative treatment.

It is a fact, though, that C1M0 patients have a better survival than C1M1 patients. Currently, there is no level-1 evidence for specific treatment of C1M0 patients, why further research is required to approach this patient group in the most comprehensive way. The focus group of our study is therefore C1M0 patients, because of the difference in opinions. Furthermore most evidence is based on gastric carcinomas, why GEJ-cancer patients are the group, we will examine.

Purpose:

Peritoneal washing cytology (PWC) is performed as a standard prediagnostic modality at Rigshospitalet, for patients with gastric- and GEJ cancer, considered resectable at preceding multidisciplinary conference. Most studies in the past 20-years have focused on gastric cancer, and not specifically GEJ-cancer.

This study will determine the usefulness of peritoneal washing cytology, and thereby verifying our own standard regarding GEJ-cancer. Furthermore, we will determine the effect of neoadjuvant chemotherapy on free peritoneal tumor cells and its correlation with overall survival.

This study is intended as a validation of our own standard.

DETAILED DESCRIPTION:
1. Background:

   The prevalence of gastroesophageal-junction cancer is increasing in Denmark with more than 400 patients per year. The 5-year overall survival is less than 10% for the 2/3 of the patients, which are not considered resectable. Even for the 1/3, which is treated with surgical intervention and neoadjuvant chemotherapy, the overall-survival is approximately 30%.

   The current Danish intended curative treatment consist of esophagectomy a.m. Ivor Lewis with extended lymphadenectomy in the abdomen and thorax. Furthermore, perioperative chemotherapy consists of 6 series neoadjuvant chemotherapy.

   Unresectable patients receive palliative chemotherapy and no resection.

   Peritoneal washing cytology is a recommended prediagnostic modality in gastric cancer. The method is used to detect free peritoneal cancer cells in the abdominal cavity, even when macroscopic carcinomatosis is not present.

   Carcinomatosis can be found in up to 19% in gastric cancer patients, often in the peritoneum. Positive peritoneal cytology (C1) can be identified in up to 7% of gastric cancer patients without metastases (C1M0). Lots of studies indicate that C1-disease is an independent prognostic predictor for decreased survival, and increased recurrence rate, comparable with M1 patients (i.e. patients with distant metastases).

   The American Joint Committee on cancer recommends that C1 patients should be treated non-surgically - even when M1 disease is not identified.

   On the basis of the above, PWC can be used to identify patients at greater risk for recurrence, and thereby not candidates for intended curative treatment.

   It is a fact, though, that C1M0 patients have a better survival than C1M1 patients. Currently, there is no level-1 evidence supporting specific treatment of C1M0 patients, why further research is required to approach this patient group in the most comprehensive way. Therefore, the focus group of our study is C1M0 patients, because of the differences in opinions. Furthermore, most evidence is based on gastric carcinomas, why GEJ-cancer patients are the group, we will examine.

   Results from other investigators regarding treatment of C1M0 patients:

   Lee et al. found a median survival of 21 months and 4 months in gastrectomized versus non-gastrectomized patients. Lorentzen et al. found a median 5-year survival of 71,4% and 25% in gastrectomized patients, who had C1 at staging laparoscopy and converted after preoperative chemotherapy versus persistent C1-disease after preoperative chemotherapy.

   Another interesting treatment modality for C1M0 patients is extensive intraperitoneal lavage (EIPL) examined by a Japanese study group. 88 C1M0 patients were randomized into three group; 1. Gastrectomy only, 2. Gastrectomy + intraperitoneal chemotherapy (IPC), and 3. Gastrectomy + IPC + EIPL. Group 3 compared to group 2 had a significant better 5 year overall survival of 43,8% versus 4,6% (p<0,0001).

   Further research is required to establish specific guideline for C1M0 patients.
2. Purpose:

   Peritoneal washing cytology (PWC) is performed as a standard prediagnostic modality at Rigshospitalet for patients, with gastric- and GEJ cancer, considered resectable at preceding multidisciplinary conference. Most studies in the past 20-years have focused on gastric cancer, and not specifically GEJ-cancer.

   This study will determine the usefulness of peritoneal washing cytology, and thereby, verify our own standard regarding GEJ-cancer. Furthermore, we will determine the effect of neoadjuvant chemotherapy on free peritoneal tumor cells, correlated with overall survival.

   See outcome measures for more detailed description. This study is intended as a validation of our own standard.
3. Methods

   Our current algorithm includes peritoneal washings performed at two different time points:

   A. Staging laparoscopy using one port technique

   o After pneumoperitoneum and oversight of the abdomen is established, a puncture is created subhepatically in the midclavicular line with a pigtail catheter ch. 10.
   * 500ml of sterile 37°C NaCl is injected through the catheter and manually dispersed throughout the abdomen by positioning the operating table in different positions.
   * At least 200ml of fluid is aspirated subhepatically through the catheter.
   * 100ml is analysed by an experienced pathologist for any malignant cancer cells.

   B. Initially, before operation (transthoracic esophagectomy): either open operation or robot assisted o Robot assisted: same technique as above o Open operation: • After abdominal incision and exploration 500ml °C of sterile NaCl is manually dispersed in the abdominal cavity.
   * Peritoneal washings is aspirated subhepatically
   * Further algorithm as described above
4. Recruiting of patients:

90 consecutive patients with biopsy verified GEJ-cancer will be included. Because PWC is already a standard guideline for this group of patients at Rigshospitalet, there will be no direct inclusion of patients.

5. Study design: Prospective feasibility study. Patients considered candidates for intented curative therapy, according to The Danish Esophagus-,GEJ- and Gastric Cancer Association (DECV), is included. Furthermore, patients must have undergone evaluation of a multidisciplinary panel of specialist including the specialties surgical gastroenterology, thoracic surgery, oncology, pathology, radiology, and clinical nuclear medicine.

6. Data: Patient data will be obtained from internal systems of Rigshospitalet including OPUS, LABKA, PatologiWEB, and ORBIT.

The following preoperative data will be obtained:

- age, sex, initial symptoms, tumour staging (TNM version 7) and histology characteristics, disease anamnesis, chemotherapy treatment, medicine anamnesis, comorbidity, postoperative complications, mortality, specifics regarding PWC such as injected volume of NaCl, procedure time, aspirated amount of fluid, and cytology findings.

7. Approval: Authorization of data retreatment is approved by The Danish Data Protection Agency.

Approval of The Danish Ethics Committee has not been applied, because the study is a validation of our own standard guideline.

8. Finances:

The following contributors have financed the study:

The Danish Cancer Society Research Center, Mogens Andreasen Fonden, Familien Erichsens familiefond, and Rigshospitalet.

All expenses have been covered.

9. Results Both negative and positive results will be published in a national and/or international journal.

10. Practical feasibility The relevant patients and the medical expertise are to find at the surgical gastroenterology department of Rigshospitalet. 120 staging laparoscopies are being performed per year in the handling of gastric cancer patients. Persons and departments involved in the study have agreed to allocate time and resources to the study. Furthermore, our department has a technician affiliated with our institution on full time basis, who is going to provide development, optimization, and assistance of projects associated with GEJ-cancer.

ELIGIBILITY:
Inclusion Criteria:

* patients with biopsy verified GEJ-cancer referred to the department of surgical gastroenterology, Rigshospitalet, which is considered resectable at MDT-conference.
* >18 years old
* informed consent

Exclusion Criteria:

* < 18 years old
* Not informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with biopsy verified GEJ-cancer referred from peripheral hospitals in the region of Sjælland and the Capitol.
  (The treatment of GEJ-cancer is centered at Rigshospitalet. All of our patients are referred from other hospitals)
Sampling Method: Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2014-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
The effect of neoadjuvant chemotherapy (NAC) on free peritoneal cancer cells (FPCCs) | 1 year
  Peritoneal washings will be performed at two time points. The first at the time of staging laparoscopy and the second initially before esophagectomy. Thereby, we will gain a measure for the effect of NAC on FPCC.
  We are interested in the following:
  * patients converting from positive cytology at staging laparoscopy to negative before surgery or reverse.
  * patients with persisting negative cytology at both measure points or persisting positive.
  These measurements for these 4 groups will be correlated with overall survival (up to 5 years).

SECONDARY OUTCOMES:
Postoperative complications | 2 weeks after surgery
  Minor complications:
  atelectasis, pleural effusion, pneumonia, chylothorax, pulmonary embolism, pneumothorax, empyema, wound infection, supraventricular arrhythmia, radiographic anastomotic leakage
  Severe complications:
  Respiratory insufficiency requiring reintubation, heart failure, cerebrovascular incidents, renal insufficiency, AMI, sepsis, death
Overall survival | up to 5 years
  Overall survival will be determined after 5 years postoperatively. In the meantime, we will assess survival after 1,2,3,4 and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Lars Bo Svendsen, Prof., MD., DMSc., Study Director — Department of surgical gastroenterology, Rigshospitalet; Michael Patrick Achiam, MD. phD., Study Chair — Department of surgical gastroenterology, Rigshospitalet; Rune Broni Strandby, Junior researcher, Principal Investigator — Department of surgical gastroenterology, Rigshospitalet
Locations (1):
- Department of surgical gastroenterology, Rigshospitalet, Copenhagen, Kbh Ø, Denmark